CLINICAL TRIAL: NCT06869291
Title: Observation of the Effect and Mechanism of Multi Tunnel Minimally Invasive Treatment for Xanthelasma Palpebrarum
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fuzhou First General Hospital Skin Disease Prevention and Control Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FZSPFY
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Xanthelasma Palpebrarum
Keywords: Xanthelasma Palpebrarum
MeSH Terms: conditions — Xanthomatosis | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Heparin Sodium Injection (Active Comparator): 1. Disinfect the area within 1cm outside the edge of the eyelid xanthoma and lesion using iodine and cotton swabs three times;
  2. Prepare heparin sodium and lidocaine in ratios of 1:1, and prepare 0.1ml of liquid per 1cm2 of lesion area;
  3. Use a 1ml syringe to insert the needle from the edge of the lesion near the eyebrow, so that it will not cover the field of view with gauze after injection;
  4. The injection depth is the gap between the epidermal layer and the dermis layer, forming an "orange peel appearance" after injection, and completely covering the lesion area;
  5. Cover the injection site with gauze and maintain for 6-8 hours.
  Interventions: Procedure: Heparin Sodium Injection
- Multi Level and Multi Tunnel Puncture Treatment (Experimental): 1. Disinfect the area within 1cm outside the edge of the eyelid xanthoma and lesion using iodine and cotton swabs three times;
  2. Use a 1ml syringe to extract lidocaine for local anesthesia of the eyelid xanthoma lesion area;
  3. Use a 1ml syringe to puncture the area between the epidermis and dermis layers, nipple layer, and reticular layer of the lesion, with the puncture endpoint at the edge of the lesion. Be careful not to penetrate the skin as much as possible, and when withdrawing the syringe, do not let the needle completely leave the puncture hole, leaving only one pinhole as much as possible; Within the same level, the distance between adjacent puncture tunnel ends is 1mm; Arrange the puncture tunnels staggered within adjacent levels;
  4. Cover the injection site with gauze and maintain for 6-8 hours.
  Interventions: Procedure: Multi level and multi tunnel puncture treatment
- Multi Level and Multi Tunnel Puncture Treatment + Heparin Sodium Injection (Experimental): 1. Disinfect the area within 1cm outside the edge of the eyelid xanthoma and lesion using iodine and cotton swabs three times;
  2. Prepare heparin sodium and lidocaine in ratios of 1:1, and prepare 0.1ml of liquid per 1cm2 of lesion area;
  3. Use a 1ml syringe to extract lidocaine for local anesthesia of the eyelid xanthoma lesion area;
  4. Use a 1ml syringe to puncture the area between the epidermis and dermis layers, nipple layer, and reticular layer of the lesion, with the puncture endpoint at the edge of the lesion. Be careful not to penetrate the skin as much as possible, and when withdrawing the syringe, do not let the needle completely leave the puncture hole, leaving only one pinhole as much as possible; Within the same level, the distance between adjacent puncture tunnel ends is 1mm; Arrange the puncture tunnels staggered within adjacent levels;
  5. Cover the injection site with gauze and maintain for 6-8 hours.
  Interventions: Procedure: Multi Level and Multi Tunnel Puncture Treatment + Heparin Sodium Injection

INTERVENTIONS:
Procedure: Multi level and multi tunnel puncture treatment — Multi level and multi tunnel puncture treatment steps
  1. Disinfect the area within 1cm outside the edge of the eyelid xanthoma and lesion using iodine and cotton swabs three times;
  2. Use a 1ml syringe to extract lidocaine for local anesthesia of the eyelid xanthoma lesion area;
  3. Use a 1ml syringe to puncture the area between the epidermis and dermis layers, nipple layer, and reticular layer of the lesion, with the puncture endpoint at the edge of the lesion. Be careful not to penetrate the skin as much as possible, and when withdrawing the syringe, do not let the needle completely leave the puncture hole, leaving only one pinhole as much as possible; Within the same level, the distance between adjacent puncture tunnel ends is 1mm; Arrange the puncture tunnels staggered within adjacent levels;
  4. Cover the injection site with gauze and maintain for 6-8 hours.
  Arms: Multi Level and Multi Tunnel Puncture Treatment
Procedure: Heparin Sodium Injection — (1) Disinfect the area within 1cm outside the edge of the eyelid xanthoma and lesion using iodine and cotton swabs three times; (2) Prepare heparin sodium and lidocaine in ratios of 1:1, and prepare 0.1ml of liquid per 1cm2 of lesion area; (3) Use a 1ml syringe to insert the needle from the edge of the lesion near the eyebrow, so that it will not cover the field of view with gauze after injection; (4) The injection depth is the gap between the epidermal layer and the dermis layer, forming an "orange peel appearance" after injection, and completely covering the lesion area; (5) Cover the injection site with gauze and maintain for 6-8 hours.
  Arms: Heparin Sodium Injection
Procedure: Multi Level and Multi Tunnel Puncture Treatment + Heparin Sodium Injection — (1) Disinfect the area within 1cm outside the edge of the eyelid xanthoma and lesion using iodine and cotton swabs three times; (2) Prepare heparin sodium and lidocaine in ratios of 1:1, and prepare 0.1ml of liquid per 1cm2 of lesion area; (3) Use a 1ml syringe to extract lidocaine for local anesthesia of the eyelid xanthoma lesion area; (4) Use a 1ml syringe to puncture the area between the epidermis and dermis layers, nipple layer, and reticular layer of the lesion, with the puncture endpoint at the edge of the lesion. Be careful not to penetrate the skin as much as possible, and when withdrawing the syringe, do not let the needle completely leave the puncture hole, leaving only one pinhole as much as possible; Within the same level, the distance between adjacent puncture tunnel ends is 1mm; Arrange the puncture tunnels staggered within adjacent levels; (5) Cover the injection site with gauze and maintain for 6-8 hours.
  Arms: Multi Level and Multi Tunnel Puncture Treatment + Heparin Sodium Injection

SUMMARY:
Dear research participants:

Participants will be invited to participate in a research project led by the Dermatology Prevention and Treatment Institute of Fuzhou First General Hospital (Huang Zhiyong) (15260471946). The research project is titled "New Directions in the Treatment of Xanthelasma Palpebrarum: Research on Hematoma Related Treatment Methods and Mechanisms".

Participants' participation in this study is voluntary, and this informed consent form provides participants with some information to help participants decide whether to participate in this clinical study. This study has been reviewed and approved by the Ethics Committee of the Dermatology Prevention and Treatment Hospital of Fuzhou First General Hospital. The Ethics Committee office phone number is 0591-83787173. If participants agree to join this study, please read it carefully and if participants have any questions, please raise them with the researcher responsible for the study.

Research objective:

Exploring whether multi tunnel minimally invasive treatment and heparin induced hematoma can initiate immune response through DAMP, mediate Toll like receptor activation of Th2 cells, secrete IL-4 and IL-13 to activate neutrophils and M2 macrophages, and then engulf cholesterol, triglycerides, and apolipoprotein in xanthelasma palpebrarum, ultimately leading to its disappearance.

DETAILED DESCRIPTION:
Heparin Sodium Injection Procedure:

1. Disinfect the XP and the area 1cm beyond the lesion margin three times using iodophor and cotton swabs.
2. Dilute heparin sodium with 0.9% saline to a concentration of 2500 - 5000 U/ml, preparing 0.1ml of liquid per 1cm² of lesion area.
3. Use a 1ml syringe to insert the needle near the edge of the lesion, the puncture site should preferably be close to the eyebrow, ensuring that the gauze cover post-injection does not obstruct the view.
4. The needle should reach the space between the epidermis and dermis layers, creating an "orange-peel appearance" post-injection, fully covering the lesion area.
5. Cover the injection site with gauze for 6-8 hours.
6. The treatment should be repeated every 5-14 days.

Autologous Blood Injection and Autologous Blood + Heparin Sodium Injection Procedure:

1. Draw blood from the patient's arm vein, preparing 0.1ml of liquid per 1cm² of lesion area.
2. Disinfect the XP and the area 1cm beyond the lesion margin three times using iodophor and cotton swabs.
3. Dilute heparin sodium with 0.9% saline/autologous blood to a concentration of 2500 - 5000 U/ml, preparing 0.1ml of liquid per 1cm² of lesion area.
4. Insert the needle from the edge of the lesion near the eyebrow using a 1ml syringe, ensuring that the gauze cover post-injection does not obstruct the field of view.
5. The needle should reach the space between the epidermis and dermis layers, creating an "orange-peel appearance" post-injection, fully covering the lesion area.
6. Cover the injection site with gauze for 6-8 hours.
7. The treatment should be repeated every 5-14 days (The next treatment can commence once the hematoma has completely resolved ).

Multi-Level Multi-Tunnel Puncture(MMP) and Multi-Level Multi-Tunnel Puncture(MMP) + Heparin Sodium Injection Procedure:

1. Disinfect the XP and the area 1cm beyond the lesion margin three times using iodophor and cotton swabs.
2. Use a 1ml syringe to inject lidocaine for local anesthesia in the XP lesion area.
3. Dilute heparin sodium with 0.9% saline to a concentration of 2500 - 5000 units/ml, preparing 0.1ml of liquid per 1cm² of lesion area (omit this step if using MMP treatment alone).
4. Use a 1ml syringe to insert the needle near the eyebrow edge of the lesion, ensuring that the gauze cover post-injection does not obstruct the view (omit this step if using MMP treatment alone).
5. The needle should reach the space between the epidermis and dermis layers, creating an "orange-peel appearance" post-injection , fully covering the lesion area (omit this step if using MMP treatment alone).
6. Use a 1ml syringe to puncture between the epidermis and dermis, within the papillary and reticular layers, with the puncture endpoint at the lesion margin. Avoid penetrating the skin completely and try to leave only one needle hole upon withdrawal. The distance between adjacent tunnel endpoints within the same layer should be 1mm; stagger the tunnels in adjacent layers .
7. Cover the injection site with gauze for 6-8 hours.
8. The treatment should be repeated every 7-14 days (The next treatment can commence once the hematoma has completely resolved ).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of xanthelasma palpebrarum
* Must be able to receive heparin sodium injection and multi tunnel minimally invasive treatment

Exclusion Criteria:

* Hemophilia
* Coronary heart disease
* Myocardial infarction
* Cerebral infarction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of regression area of xanthelasma palpebrarum | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- No. 243 Xihong Road, Gulou District, Fuzhou City, Fujian Province, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No